CLINICAL TRIAL: NCT00004907
Title: High-Dose Chemoradiotherapy With Stem Cell Allogeneic Cellular Rescue in Patients With Relapsed or Refractory Hematologic Malignancy - A Phase I/II Study
Brief Title: Chemotherapy and Radiation Therapy Plus Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Relapsed or Refractory T-cell Lymphoma, Hodgkin's Lymphoma, or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: NU 95H4T; NU-95H4T; NCI-G00-1692
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Busulfan; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: etoposide
Procedure: allogeneic bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Bone marrow or peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and radiation therapy and kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of chemotherapy and radiation therapy plus bone marrow or peripheral stem cell transplantation in treating patients who have refractory or relapsed T-cell lymphoma, Hodgkin's lymphoma, or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of an intensive program of chemoradiotherapy followed by HLA identical related bone marrow or peripheral blood stem cell transplantation in patients with relapsed or refractory cutaneous T-cell lymphoma, Hodgkin's lymphoma, or non-Hodgkin's lymphoma.
* Determine the response rate and disease free survival in patients treated with this regimen.

OUTLINE: HLA identical related donors undergo harvest of bone marrow or peripheral blood stem cells (PBSC).

Patients are assigned to one of two treatment groups based on prior radiation to abdomen or mediastinum:

* Group A (prior radiation no greater than 2,000 cGy): Patients with complete response (CR) or partial response (PR) after completion of chemotherapy receive cyclophosphamide IV over 1 hour on days -6 and -5, followed by total body irradiation twice daily on days -4 to -1. Patients with minimal response after completion of chemotherapy receive cyclophosphamide IV over 1 hour on days -8 and -7, followed by etoposide IV over 30 hours beginning on day -6, followed by total body irradiation twice daily on days -4 to -1.
* Group B (prior radiation greater than 2,000 cGy): Patients with CR or PR after completion of chemotherapy receive oral busulfan every 6 hours on days -7 to -4, followed by cyclophosphamide IV over 1 hour on days -3 and -2. Patients with minimal response after completion of chemotherapy receive oral busulfan every 6 hours on days -9 to -6, followed by cyclophosphamide IV over 1 hour on days -5 and -4, followed by etoposide IV over 30 hours beginning on day -3.
* Both groups: Bone marrow or PBSC are reinfused on day 0. Patients with bulky nodal disease (greater than 5 cm) may undergo involved field radiotherapy two weeks before transplantation.

Patients are followed every month for 1 year.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven relapsed or refractory cutaneous T-cell lymphoma, Hodgkin's lymphoma, or non-Hodgkin's lymphoma of the following types:

  * Diffuse small lymphocytic/marginal zone
  * Grade I follicular small cleaved cell
  * Grade II follicular mixed cell
  * Diffuse small cleaved cell
  * Grade III follicular large cell
  * Diffuse mixed cell
  * Diffuse large cell
  * Immunoblastic large cell
* HLA identical related donor available

  * Phenotypically HLA identical, MLC nonstimulatory donor eligible if no HLA identical related donor is available
* Relapse following autologous bone marrow transplantation allowed if an HLA identical related donor is available
* Eligible for total body irradiation
* No active uncontrolled CNS disease NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* Over 15 to physiologic age 60

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No congestive heart failure
* No myocardial infarction within the past 3 months
* No significant arrhythmia requiring medication
* Resting LVEF normal

Pulmonary:

* No significant nonneoplastic pulmonary disease (e.g., chronic obstructive pulmonary disease) that would preclude therapy with cytotoxic drugs
* DLCO at least 50% of predicted* OR
* FEV1 and/or FVC at least 50% of predicted* NOTE: * Unless due to lymphoma, including Hodgkin's lymphoma

Other:

* Not pregnant
* Negative pregnancy test
* No active serious medical condition that would preclude aggressive cytotoxic chemotherapy
* HIV negative and no clinical evidence of AIDS

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-10; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo I. Gordon, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States